CLINICAL TRIAL: NCT03262935
Title: A Multi-centre, Open-label, Randomized Clinical Trial Comparing the Efficacy and Safety of the Antibody-drug Conjugate SYD985 to Physician's Choice in Patients With HER2-positive Unresectable Locally Advanced or Metastatic Breast Cancer
Brief Title: SYD985 vs. Physician's Choice in Participants With HER2-positive Locally Advanced or Metastatic Breast Cancer
Acronym: TULIP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Byondis B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYD985.002
Record Dates: First submitted 2017-08-16; First posted 2017-08-25 (Actual); Results first posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-06

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — trastuzumab duocarmazine; Lapatinib; CCAAT-Enhancer-Binding Protein-beta; Capecitabine; Capsules; Trastuzumab; Vinorelbine; eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- (vic-)trastuzumab duocarmazine (Experimental): SYD985, every 3 weeks (Q3W)
  Interventions: Drug: (vic-)trastuzumab duocarmazine
- Physician's choice (Active Comparator): 1. Lap/Cap
  2. T/Cap
  3. T/Vino
  4. T/Eri
  Interventions: Drug: Physician's choice

INTERVENTIONS:
Drug: (vic-)trastuzumab duocarmazine — Intravenous SYD985, Q3W
  Other Names: SYD985; Trastuzumab vc-seco-DUBA
  Arms: (vic-)trastuzumab duocarmazine
Drug: Physician's choice — See drug label
  Other Names: Lapatinib (Lap); Capecitabine (Cap); Trastuzumab (T); Vinorelbine (Vino); Eribulin (Eri)
  Arms: Physician's choice

SUMMARY:
The purpose of this study is to demonstrate that SYD985 [(vic-)trastuzumab duocarmazine] is superior to physician's choice in prolonging progression free survival.

DETAILED DESCRIPTION:
This study is designed as a randomized, active-controlled, superiority study in patients with unresectable locally advanced or metastatic HER2-positive breast cancer. The patients should have had either progression during or after at least two HER2-targeting treatment regimens for locally advanced or metastatic disease or progression during or after (ado-)trastuzumab emtansine treatment.

Eligible patients will be randomly assigned (2:1) to receive SYD985 or physician's choice treatment until disease progression, unacceptable toxicity or study termination by the Sponsor. During treatment, patients will have to visit the clinical site to assess efficacy, quality of life (QoL), and safety using standardized criteria.

ELIGIBILITY:
Main Inclusion Criteria:

* Female patients with histologically-confirmed, unresectable locally advanced or metastatic breast cancer;
* Patients should have had either progression during or after at least two HER2-targeting treatment regimens for locally advanced or metastatic disease or progression during or after (ado-)trastuzumab emtansine treatment for locally advanced or metastatic disease;
* HER2-positive tumor status;
* Patients must have measurable or non-measurable disease that is evaluable per RECIST 1.1;
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2;
* Estimated life expectancy > 12 weeks at randomization;
* Adequate organ function and blood cell counts.

Main Exclusion Criteria:

* Current or previous use of a prohibited medication as listed in the protocol;
* History of infusion-related reactions and/or hypersensitivity to trastuzumab, (ado-)trastuzumab emtansine;
* History of keratitis;
* Severe, uncontrolled systemic disease at screening;
* Left Ventricular Ejection Fraction (LVEF) < 50%, or a history of clinically significant decrease in LVEF during previous treatment with trastuzumab or (ado-)trastuzumab emtansine;
* Cardiac troponin value above the Upper Limit of Normal (ULN);
* History of clinically significant cardiovascular disease;
* Untreated brain metastases, symptomatic brain metastases, brain metastases requiring steroids to manage symptoms, or treatment for brain metastases within 8 weeks prior to randomization;
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 437 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evelyn van den Tweel, PhD, Study Director — Byondis B.V., The Netherlands
Locations (90):
- United States (23):
  - Southern Cancer Center, Mobile, Alabama
  - Arizona Clinical Research Center, Tucson, Arizona
  - Moores UCSD Cancer Center, San Diego, California
  - Woodlands Medical Specialists, Pensacola, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Cancer Center of Kansas, Wichita, Kansas
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - FirstHealth Outpatient Cancer Center, Pinehurst, North Carolina
  - Toledo Clinic Cancer Center, Toledo, Ohio
  - Northwest Cancer Specialists, Portland, Oregon
  - Magee-Womens Hospital of UPMS, Pittsburgh, Pennsylvania
  - Texas Oncology PA (Texas Oncology-Dallas Presbyterian Hospital), Dallas, Texas
  - Texas Oncology- Baylor Charles A. Sammor, Dallas, Texas
  - Texas Oncology - Denton South, Denton, Texas
  - Texas Oncology-Memorial City, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Texas Oncology-San Antonio Northeast, San Antonio, Texas
  - Texas Oncology-Tyler, Tyler, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
- Belgium (7):
  - Institut Jules Bordet, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - University Hospital Antwerp, Edegem
  - UZ Gent, Ghent
  - AZ Groeninge, Kortrijk
  - UZ Leuven - campus Gasthuisberg, Leuven
  - CHU Liege, Liège
- Canada (4):
  - Cross Cancer Institute, Edmonton
  - BC Cancer Agency Centre for the Southern Interior, Kelowna
  - McGill University Health Centre, Montreal
  - The Ottawa Hospital Cancer Center, Ottawa
- Denmark (3):
  - Sealand University Hospital, Næstved
  - Odense University Hospital, Odense
  - Sønderborg sygehus, Sønderborg
- France (12):
  - Institut de Cancerologie de l'ouest, Angers
  - Institut Bergonie, Bordeaux
  - CH Fleyrait, Bourg-en-Bresse
  - Centre Hospitalier Lyon Sud, Corbeil-Essonnes
  - Centre Georges francois leclerc, Dijon
  - Oscar Lambret, Lille
  - CHR Metz-Thionville, Metz
  - Hopital Prive du Confluent, Nantes
  - Hopital Saint Louis, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Henri Becquere, Rouen
  - Centre Paul Strauss, Strasbourg
- Italy (14):
  - IRCCS Istituto Oncologico, Bari
  - Policlinico S.Orsola-Malpighi, Bologna
  - Azienda Ospedaliera Garibaldi- Nesima, Catania
  - Azienda Ospedaliero - Universitaria Careggi, Florence
  - IRCCS Ospedale San Raffaele, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Europeo di Oncologia, Milan
  - University Hospital of Modena, Modena
  - Ospedale San Gerardo-Asst Monza, Monza
  - Istituto Oncologico Veneto Irccs, Padua
  - Nuovo Ospedale Santo Stefano, Prato
  - Istituto Nazionale dei Tumori Regina Elena, Roma
  - Azienda Ospedaliera Sant'Andrea, Roma
  - Casa Sollievo Della Sofferenza, San Giovanni Rotondo
- Netherlands (3):
  - Radboud University Medical Center, Nijmegen, Gelderland
  - VU Medical Center, Amsterdam, North Holland
  - University Medical Center Groningen, Groningen
- Singapore (2):
  - National University Cancer Institute, Singapore
  - National Cancer Centre Singapore, Singapore
- Spain (11):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Quironsalud, Barcelona
  - Hospital Universitari Vall d'Hebron Vall d' Hebron Institute of Oncology (VHIO), Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Institut Catala D'oncologia, Barcelona
  - Hospital Arnau de Vilanova, Lleida
  - Hospital General Universitario Gregorio Marañón, Madrid
  - IOB del Hospital Ruber Internacional, Madrid
  - Hospital HM Universitario Sanchinarro, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Sweden (4):
  - Gävle Sjukhus Onkologkliniken, Gävle
  - Sahlgrenska University Hospital, Gothenburg
  - Karolina University Hospital, Stockholm
  - Akademiska Hospital, Uppsala
- United Kingdom (7):
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Bebington
  - Velindre Cancer Centre VCC, Cardiff
  - Beatson West of Scotland Cancer Centre, Glasgow
  - The Royal Marsden NHS Foundation Trust, London
  - SCRI UK, London
  - The Christie NHS Foundation, Manchester
  - Oxford University NHS hospital, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Turner N, Saura C, Aftimos P, van den Tweel E, Oesterholt M, Koper N, Colleoni M, Kaczmarek E, Punie K, Song X, Armstrong A, Bianchi G, Stradella A, Ladoire S, Lim JSJ, Quenel-Tueux N, Tan TJ, Escriva-de-Romani S, O'Shaughnessy J; TULIP Trial Investigators. Trastuzumab Duocarmazine in Pretreated Human Epidermal Growth Factor Receptor 2-Positive Advanced or Metastatic Breast Cancer: An Open-Label, Randomized, Phase III Trial (TULIP). J Clin Oncol. 2025 Feb 10;43(5):513-523. doi: 10.1200/JCO.24.00529. Epub 2024 Oct 23. PMID 39442070

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 751 participants were screened, out of which, 437 participants were randomized into the study.
Groups:
- Physician's Choice: 1. Lap/Cap
  2. T/Cap
  3. T/Vino
  4. T/Eri
  Physician's choice: See drug label
Period: Overall Study
Arm/Group | (Vic-)Trastuzumab Duocarmazine | Physician's Choice
Started | 291 | 146
Completed | 0 | 0
Not Completed | 291 | 146
Not completed — Withdrawal by Subject | 6 | 7
Not completed — End Of Follow Up By Sponsor | 90 | 41
Not completed — Death | 181 | 94
Not completed — Lost to Follow-up | 9 | 4
Not completed — Other reason | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | (Vic-)Trastuzumab Duocarmazine | Physician's Choice | Total
Number analyzed (Participants) | 291 | 146 | 437
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (11.2) | 57.3 (10.97) | 56.4 (11.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 291 | 146 | 437
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 8 | 19
  Not Hispanic or Latino | 225 | 103 | 328
  Unknown or Not Reported | 55 | 35 | 90
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 29 | 17 | 46
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 202 | 95 | 297
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 55 | 32 | 87
Region of Enrollment [Number; unit: participants]
  Canada | 15 | 9 | 24
  Netherlands | 3 | 0 | 3
  Sweden | 4 | 4 | 8
  Singapore | 20 | 15 | 35
  Belgium | 25 | 15 | 40
  United States | 34 | 19 | 53
  Denmark | 7 | 3 | 10
  Italy | 50 | 20 | 70
  United Kingdom | 43 | 16 | 59
  France | 46 | 22 | 68
  Spain | 44 | 23 | 67
BMI [Mean (Standard Deviation); unit: kg/m2] — Population: The number analyzed differs from the overall because height was missing for 3 patients in the SYD985 group and for 1 patient in the Physician's choice group.
  kg/m2
    number analyzed (Participants) | 288 | 145 | 433
    (all) | 25.14 (5.0) | 25.54 (6.1) | 25.28 (5.4)
Childbearing potential [Count of Participants; unit: Participants]
  Yes | 64 | 32 | 96
  No - postmenopausal | 204 | 105 | 309
  No - surgically sterilized | 23 | 9 | 32

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression-free survival is defined as the time from the date of randomization to the date of first documented disease progression by central assessment according to Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 or death due to any cause, whichever occurred earlier.
Time Frame: baseline until primary analysis data cut-off date of 31March2021
Population: Full-analysis set (FAS) was used for this primary endpoint analysis. FAS comprises all randomized patients, which were analyzed according to the treatment group and strata they have been assigned to during the randomization procedure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | (Vic-)Trastuzumab Duocarmazine | Physician's Choice
Number analyzed (Participants) | 291 | 146
months | 7.0 [5.4 to 7.2] | 4.9 [4.0 to 5.5]
Statistical Analysis 1: Comparison: (Vic-)Trastuzumab Duocarmazine vs Physician's Choice; A stratified Cox regression analysis was used to estimate the hazard ratio of PFS, along with 95% CIs. Stratification factors assigned at randomization were world region (Europe, Singapore, and North America), number of prior treatment lines for locally advanced or metastatic breast cancer (excluding hormone therapy) (1 to 2, >2), and prior treatment with pertuzumab (yes, no); Test type: Superiority; p = 0.002, Log Rank — P-value from stratified log-rank test for median estimate of PFS: stratified according to the randomization stratification factors; Hazard Ratio (HR) = 0.6401, 95% CI 2-sided [0.4885 to 0.8389]

2. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from date of randomization to death due to any cause.
Time Frame: baseline until final Overall Survival analysis data cut-off date of 30June2022
Population: Full-analysis set (FAS) was used for the overall survival analysis. FAS comprises all randomized patients, which were analyzed according to the treatment group and strata they have been assigned to during the randomization procedure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | (Vic-)Trastuzumab Duocarmazine | Physician's Choice
Number analyzed (Participants) | 291 | 146
months | 21.0 [18.1 to 25.0] | 19.5 [14.2 to 23.1]
Statistical Analysis 1: Comparison: (Vic-)Trastuzumab Duocarmazine vs Physician's Choice; A stratified Cox regression analysis was used to estimate the hazard ratio of OS, along with 95% CIs. Stratification factors assigned at randomization were world region (Europe, Singapore, and North America), number of prior treatment lines for locally advanced or metastatic breast cancer (excluding hormone therapy) (1 to 2, >2), and prior treatment with pertuzumab (yes, no); Test type: Superiority; p = 0.236, Log Rank — P-value from stratified log-rank test for Kaplan-Meier estimate of median OS: stratified according to the randomization stratification factors; Hazard Ratio (HR) = 0.868, 95% CI 2-sided [0.676 to 1.1145]

3. Secondary Outcome: Objective Response Rate
Description: Objective Response Rate is defined as the proportion of patients with a centrally assessed best overall response of complete response or partial response according to RECIST v1.1.
Time Frame: baseline until primary analysis data cut-off date of 31March2021
Population: Full-analysis set (FAS) was used for this primary endpoint analysis. FAS comprises all randomized patients, which were analyzed according to the treatment group and strata they have been assigned to during the randomization procedure. Only patients with measurable disease at baseline were included in the analysis of ORR.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | (Vic-)Trastuzumab Duocarmazine | Physician's Choice
Number analyzed (Participants) | 252 | 122
percentage of patients | 27.8 [22.3 to 33.7] | 29.5 [21.6 to 38.4]
Statistical Analysis 1: Comparison: (Vic-)Trastuzumab Duocarmazine vs Physician's Choice; The Cochran-Mantel-Haenszel test (strata based on the baseline stratification factors) was used to compare the two treatment groups with respect to the ORR at two-sided 5% level of significance; Test type: Superiority; p = 0.732, Cochran-Mantel-Haenszel — P-value from Cochran-Mantel-Haenszel test including the randomization stratification factors

4. Secondary Outcome: Investigator Assessed Progression Free Survival
Description: Progression-free survival is defined as the time from the date of randomization to the date of first documented disease progression by investigator assessment according to RECIST v1.1 or death due to any cause, whichever occurred earlier.
Time Frame: baseline until primary analysis data cut-off date of 31March2021
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | (Vic-)Trastuzumab Duocarmazine | Physician's Choice
Number analyzed (Participants) | 291 | 146
months | 6.9 [6.0 to 7.2] | 4.6 [4.0 to 5.6]
Statistical Analysis 1: Comparison: (Vic-)Trastuzumab Duocarmazine vs Physician's Choice; A stratified Cox regression analysis was used to estimate the HR of PFS, along with the 95% CI. The treatment groups were compared using the 2-sided stratified log-rank test; Test type: Superiority; p < 0.001, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.5995, 95% CI 2-sided [0.4666 to 0.7703]

5. Secondary Outcome: Patient Reported Outcomes for Health Related Quality of Life
Description: Change in the global health status/Quality of Life (QoL) scale score of the European Organization for Research and Treatment for Cancer (EORTC) Quality of Life Questionnaire C30 from baseline (cycle 1). The raw score (1 to 7) has been transformed to a score ranging from 0 to 100. A higher score means a better outcome: hence a positive change from baseline means an improvement in global health status/Quality of Life and a negative change from baseline means a worsening of global health status/Quality of Life.
Time Frame: baseline until primary analysis data cut-off date of 31March2021
Population: Full-analysis set (FAS) was used for the overall survival analysis. FAS comprises all randomized patients, which were analyzed according to the treatment group and strata they have been assigned to during the randomization procedure. Here, 'Number analyzed' = participants with available QoL for each specified cycle.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | (Vic-)Trastuzumab Duocarmazine | Physician's Choice
Number analyzed (Participants) | 291 | 146
scores on a scale
  Cycle 2: number analyzed (Participants) | 222 | 95
  Cycle 2 | 0.17 [-2.70 to 3.04] | -3.88 [-7.79 to 0.03]
  Cycle 3: number analyzed (Participants) | 195 | 89
  Cycle 3 | -1.88 [-4.83 to 1.07] | -2.99 [-7.00 to 1.02]
  Cycle 4: number analyzed (Participants) | 190 | 79
  Cycle 4 | -2.48 [-5.46 to 0.50] | -9.01 [-13.23 to -4.80]
  Cycle 5: number analyzed (Participants) | 154 | 63
  Cycle 5 | -2.51 [-5.69 to 0.67] | -5.77 [-10.34 to -1.21]
  Cycle 7: number analyzed (Participants) | 114 | 47
  Cycle 7 | -5.65 [-9.19 to -2.10] | -6.75 [-11.92 to -1.58]
  Cycle 9: number analyzed (Participants) | 78 | 31
  Cycle 9 | -8.14 [-12.27 to -4.02] | -11.25 [-17.41 to -5.09]
  Cycle 11: number analyzed (Participants) | 51 | 19
  Cycle 11 | -10.70 [-15.66 to -5.75] | -10.38 [-18.08 to -2.69]
  Cycle 13: number analyzed (Participants) | 26 | 15
  Cycle 13 | -13.40 [-20.31 to -6.48] | -12.89 [-21.33 to -4.45]
  Cycle 15: number analyzed (Participants) | 16 | 12
  Cycle 15 | -11.90 [-20.41 to -3.39] | -14.12 [-23.91 to -4.33]
  Cycle 17: number analyzed (Participants) | 12 | 7
  Cycle 17 | -4.31 [-14.48 to 5.86] | -0.71 [-13.26 to 11.83]
  Cycle 19: number analyzed (Participants) | 6 | 4
  Cycle 19 | -5.45 [-21.05 to 10.16] | 1.66 [-13.84 to 17.16]
  Cycle 21: number analyzed (Participants) | 4 | 5
  Cycle 21 | 11.68 [-9.76 to 33.12] | -11.23 [-26.16 to 3.71]
  Cycle 23: number analyzed (Participants) | 2 | 2
  Cycle 23 | 5.30 [-26.04 to 36.65] | -7.00 [-29.18 to 15.17]
  Cycle 25: number analyzed (Participants) | 1 | 1
  Cycle 25 | 18.76 [-14.63 to 52.16] | -11.48 [-42.96 to 19.99]
  Cycle 27: number analyzed (Participants) | 2 | 1
  Cycle 27 | 0.49 [-33.40 to 34.37] | -5.41 [-38.83 to 28.02]
  Cycle 29: number analyzed (Participants) | 0 | 1
  Cycle 29 |  | -6.54 [-40.45 to 27.37]
  Cycle 33: number analyzed (Participants) | 0 | 1
  Cycle 33 |  | -7.11 [-41.14 to 26.92]
  Cycle 35: number analyzed (Participants) | 0 | 1
  Cycle 35 |  | -15.73 [-49.79 to 18.33]
Statistical Analysis 1: Comparison: (Vic-)Trastuzumab Duocarmazine vs Physician's Choice; The change from baseline in the global health status/QoL scale transformed score was analyzed using a mixed model repeated measurement (MMRM) approach; Test type: Superiority; p = 0.473, MMRM

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from signing of the ICF up to the treatment discontinuation visit. The safety data reported here is based on data collected up to the data cut off date of 31 March 2021.
Arm/Group | (Vic-)Trastuzumab Duocarmazine | Physician's Choice
All-Cause Mortality (participants affected / at risk) | 181/288 | 94/137
Serious Adverse Events (participants affected / at risk) | 53/288 | 12/137
Other Adverse Events (participants affected / at risk) | 278/288 | 132/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | (Vic-)Trastuzumab Duocarmazine (N=288) | Physician's Choice (N=137)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Haemorrhagic tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 0 (0)
Drug intolerance (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 2 (3) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
Staphylococcus test positive (Investigations) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (5) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 2 (3) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Eyelid ptosis (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (2) | 0 (0)
Livedo reticularis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (5) | 1 (1)
Wound infection (Infections and infestations) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (2) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (2)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | (Vic-)Trastuzumab Duocarmazine (N=288) | Physician's Choice (N=137)
Weight decreased (Investigations) | 29 (45) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 16 (26) | 10 (14)
Platelet count decreased (Investigations) | 16 (28) | 0 (0)
Neutrophil count decreased (Investigations) | 14 (25) | 14 (26)
Alanine aminotransferase increased (Investigations) | 12 (19) | 10 (17)
Headache (Nervous system disorders) | 33 (37) | 16 (23)
Dysgeusia (Nervous system disorders) | 22 (26) | 4 (5)
Dizziness (Nervous system disorders) | 21 (22) | 7 (7)
Neuropathy peripheral (Nervous system disorders) | 16 (29) | 8 (16)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (7) | 7 (11)
Fatigue (General disorders) | 96 (162) | 41 (66)
Asthenia (General disorders) | 58 (91) | 23 (34)
Pyrexia (General disorders) | 23 (26) | 13 (15)
Oedema peripheral (General disorders) | 22 (30) | 3 (4)
Mucosal inflammation (General disorders) | 17 (20) | 8 (10)
Anaemia (Blood and lymphatic system disorders) | 41 (85) | 17 (35)
Neutropenia (Blood and lymphatic system disorders) | 31 (75) | 33 (76)
Thrombocytopenia (Blood and lymphatic system disorders) | 17 (23) | 7 (13)
Conjunctivitis (Eye disorders) | 110 (218) | 3 (3)
Keratitis (Eye disorders) | 110 (202) | 11 (11)
Dry eye (Eye disorders) | 87 (117) | 14 (15)
Lacrimation increased (Eye disorders) | 53 (74) | 2 (2)
Blepharitis (Eye disorders) | 36 (53) | 2 (2)
Punctate keratitis (Eye disorders) | 32 (45) | 3 (4)
Vision blurred (Eye disorders) | 23 (30) | 1 (1)
Periorbital oedema (Eye disorders) | 17 (29) | 0 (0)
Nausea (Gastrointestinal disorders) | 73 (103) | 43 (64)
Diarrhoea (Gastrointestinal disorders) | 60 (82) | 49 (92)
Constipation (Gastrointestinal disorders) | 52 (74) | 24 (28)
Vomiting (Gastrointestinal disorders) | 36 (52) | 23 (37)
Dry mouth (Gastrointestinal disorders) | 26 (28) | 6 (6)
Stomatitis (Gastrointestinal disorders) | 24 (34) | 17 (17)
Abdominal pain (Gastrointestinal disorders) | 19 (30) | 11 (17)
Abdominal pain upper (Gastrointestinal disorders) | 18 (20) | 9 (12)
Dyspepsia (Gastrointestinal disorders) | 13 (15) | 9 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 48 (60) | 14 (17)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 42 (52) | 17 (27)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 19 (23) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14 (17) | 8 (9)
Alopecia (Skin and subcutaneous tissue disorders) | 62 (74) | 16 (21)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 32 (36) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 27 (27) | 8 (8)
Rash (Skin and subcutaneous tissue disorders) | 17 (18) | 5 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 15 (16) | 2 (2)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 32 (70)
Insomnia (Psychiatric disorders) | 23 (24) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 31 (36) | 11 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 22 (23) | 11 (14)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 (20) | 12 (19)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (14) | 7 (7)
Urinary tract infection (Infections and infestations) | 25 (28) | 14 (14)
Upper respiratory tract infection (Infections and infestations) | 9 (12) | 8 (11)
Decreased appetite (Metabolism and nutrition disorders) | 61 (75) | 15 (20)
Hypokalaemia (Metabolism and nutrition disorders) | 11 (13) | 9 (12)
Hypomagnesaemia (Metabolism and nutrition disorders) | 7 (7) | 7 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI agrees to provide to the Sponsor 60 days prior to intended submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the study. The Sponsor has the right to review and comment with respect to publications, abstracts, slides, and manuscripts including the data analysis and presentation. In case of disagreement, efforts will be undertaken to resolve any such issues, but the ultimate decision remains with the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2021-01-18): https://cdn.clinicaltrials.gov/large-docs/35/NCT03262935/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-29): https://cdn.clinicaltrials.gov/large-docs/35/NCT03262935/SAP_001.pdf